CLINICAL TRIAL: NCT03916094
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Pharmacodynamics of HLX22 Monoclonal Antibody Injection (HER2 Monoclonal Antibody) in Patients With Advanced Solid Tumours Overexpressing HER2
Brief Title: Evaluate Safety, Tolerability and Pharmacokinetics of HLX22 in Patients With Advanced Solid Tumors Overexpressing HER2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX22-001
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumor
Keywords: overexpressing HER2
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX22 group (Experimental): HLX22, at four dose levels (3, 10, 25mg/kg), to be intravenously injected once every three weeks; Study drugs given until disease progression, one year of treatment, withdrawal from the study or death
  Interventions: Drug: HLX22

INTERVENTIONS:
Drug: HLX22 — Humanized Anti-Human Epidermal Growth Factor Receptor-2 Monoclonal Antibody
  Other Names: HER2 Monoclonal Antibody

SUMMARY:
a single-center, open-label, dose-escalation Phase I clinical trial to evaluate the safety and the tolerability of HLX22 in patients with advanced solid tumors overexpressing HER2 after failure of standard of care.

DETAILED DESCRIPTION:
This study is an open-label and dose escalation study aimed at exploring the safety and MTD of HLX22.

three dose levels are designed for HLX22 in this study: 3, 10, and 25 mg/kg/3 weeks. The 3 mg/kg/3 weeks will serve as the starting dose. The study will use a 3+3 design to assign doses to the patients, and thereby determine the MTD of HLX22.

ELIGIBILITY:
Inclusion Criteria:

Patients with child-bearing potential must agree to and be able to use effective contraceptive measures.

At least 28 days from prior major surgery, prior cytotoxic chemotherapy, prior hormonal therapy (except for androgen-deprivation therapy in patients with prostate cancer), prior therapy with investigational products (or medical device) or local radiotherapy, at least 42 days from prior chemotherapy with nitrosoureas or mitomycin C, and at least 42 days from prior immunotherapy before the first dose of HLX22.

At least one bi-dimensionally measurable lesion to be used as the basis for evaluation.

ECOG performance status of ≤ 1 at study entry. Patients with histologically-proven HER2-positive advanced or metastatic solid tumours who are either non-responsive or intolerant to standard therapies.

HER2-positive tumours that are confirmed by immunohistochemistry (IHC) and:

1. HER2 mutation of at least 3+ (+++) or
2. HER2 mutation of at least 2+ (++) and fluorescence in situ hybridization (FISH) test positive.

Adequate haematologic functions Adequate hepatic functions Adequate renal functions Adequate cardiac functions For patients with hepatocellular carcinoma, Child-Pugh score has to be A. Able to receive treatment and examinations as required by the study protocol. Life expectancy > 3 months. Exclusion Criteria Patients with history of alcohol or drug abuse, or positive for alcohol breath test before dosing.

Patients who still have ≥ Grade 2 toxicities from prior therapies (except for Grade 2 alopecia).

Concurrent unstable or uncontrolled medical conditions with either of the following:

* Active systemic infections requiring intravenous antibiotic;
* Poorly controlled hypertension, or poor compliance with anti-hypertensive agents;
* Clinically significant arrhythmia, unstable angina pectoris, congestive heart failure (New York Heart Association [NYHA] Grade III or IV) or acute myocardial infarction within 6 months;
* Uncontrolled diabetes mellitus or poor compliance with hypoglycemics;
* NCI CTCAE Grade ≥ 2 hypercalcemia;
* Presence of chronically unhealed wound or ulcers;
* Other chronic diseases which, in the opinion of the Investigator, may compromise the safety of the patient or the integrity of the study.

Patients with history of interstitial lung disease. Patients with newly diagnosed or symptomatic brain metastases Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix (patients with a previous malignancy but without evidence of disease for ≥ 3 years can participate).

Patients have received a cumulative dose of doxorubicin (or equivalent) of ≥ 360 mg/m2.

Patients have participated in another clinical study within 4 weeks (in the case of a clinical study of a monoclonal antibody drug, 3 months or 5 half-lives, whichever is longer) prior to the enrolment, or patients have intended to participate in another clinical study during the period of the study.

Female patients in pregnancy (confirmed by ß-HCG test) or breastfeeding. Known history of human immunodeficiency virus (HIV) infection. Patients with active hepatitis B (positive for hepatitis B core antibody [HBcAb], or hepatitis B surface antigen [HBsAg], along with hepatitis B virus [HBV] DNA titre > the limit of normal defined by the study site), or hepatitis C (positive for hepatitis C antibody).

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of HLX22 in patients with advanced solid tumors overexpressing HER2 | from day1 to day 42(cycle 1 and cycle2 ,each cycle is 21days)
  The MTD is the dose with toxicity rate (estimated by isotonic regression) most approximate to the target one (30%).

SECONDARY OUTCOMES:
the pharmacokinetic characteristics of HLX22 at different doses in patients. | cycle1 to cycle 8 ,and 28-day follow-up visit after the last infusion (if possible),(each cycle is 21 days).
  Area under the plasma concentration versus time curve (AUC) for single dose and multiple doses
the pharmacodynamic characteristics of HLX22 at different doses in patients | cycle 1 to cycle 6 (each cycle is 21 days)
  the concentration of soluble HER1 and HER2 in serum
the immunogenicity of HLX22 in humans | cycle 1 to cycle 6 (each cycle is 21 days)
  anti-HLX22 antibodies in serum

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu X, Ding Y, Wang Q, Yang G, Zhou L, Wang Q. HLX22, an anti-HER-2 monoclonal antibody, in patients with advanced solid tumors overexpressing human epidermal growth factor receptor 2: an open-label, dose-escalation, phase 1 trial. Invest New Drugs. 2023 Jun;41(3):473-482. doi: 10.1007/s10637-023-01338-7. Epub 2023 May 4. PMID 37140695